CLINICAL TRIAL: NCT03166228
Title: Hematological, Biochemical and Hemodynamic Changes During Operative Hysteroscopy Using Consecutive Distension Media
Brief Title: Hemodynamic Changes During Operative Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed sonbaty, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ahmed 2017
Record Dates: First submitted 2017-05-13; First posted 2017-05-25 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal saline0.9% (Active Comparator): 0.9% saline distension media is used as long as diathermy is not in use
  Interventions: Drug: Normal Saline 0.9% Infusion Solution Bag
- 1.5% GLYCINE (Placebo Comparator): 1.5% GLYCINE DURING OPERATIVE HYSTEROSCOPY as long as diathermy is in use
  Interventions: Drug: 1.5% Glycine only

INTERVENTIONS:
Drug: Normal Saline 0.9% Infusion Solution Bag — 0.9% saline as distension medium as long as diathermy is not in use
  Arms: normal saline0.9%
Drug: 1.5% Glycine only — 1.5% Glycine alone during hysteroscopy as long as diathermy is in use
  Arms: 1.5% GLYCINE

SUMMARY:
Hysteroscopy is a minimally invasive gynaecological procedure in which an endoscopic optical lens is inserted through the cervix into the endometrial cavity to assists in the diagnosis of a vast number of uterine pathologies Historically, urologists used the resectoscope to perform a transurethral prostatectomy. This instrument was later modified to accommodate gynaecological applications. Operative hysteroscopy became popular after improvements in endoscopic technology and instruments in the 1970s and after the introduction of fluid distension media in the 1980s (1). During the past 2 decades, hysteroscopy has been increasingly used for operative procedures

DETAILED DESCRIPTION:
Operative hysteroscopy has become a standard surgical treatment for abnormal uterine bleeding unresponsive to conservative medical management since it was shown as a safe and effective alternative to hysterectomy.(2,3) Monopolar resectoscope necessitates an irrigating fluid that should be a non-conductive and salt free solution such as glycine 1.5% or sorbitol 3%.(4) Physiologic irrigating fluids (e.g. saline 0.9%) are contraindicated with these instruments since electric current generated by any monopolar electro surgical unit is preferentially conducted through low impedance fluid rather than through tissue and consequently it's difficult to initiate cutting and impossible to create significant tissue coagulation with these devices The clinical drawback of non-conductive irrigating solution (e.g. glycine 1.5%) is the risk of excessive fluid absorption leading to symptomatic dilutional hyponatremia and for hypotonic solutions, hypo-osmolarity and secondary cerebral oedema as Glycine is metabolized to carbon dioxide, water and ammonia, and may lead to intra-cellular over hydration and neurotoxicity which is clinically reflected as hypoxemia, agitation, nausea and hypertension.(5).Although rare, irreversible neurologic damage and death have been reported after excessive absorption of salt free irrigating solutions during routine operative hysteroscopy(6)Theoretically, distension with 0.9% saline as a distension medium avoids most of the above mentioned risks associated with hyper absorption of non electrolytic distension media(7) However, there is no doubt that excessive absorption of normal saline can be fatal(8).

Recently , it has been suggested that the type of anesthesia could modify fluid absorption(9). General anaesthesia has been associated with less Glycine absorption than epidural anaesthesia: the latter being associated with systemic vasodilatation(9).

ELIGIBILITY:
Inclusion Criteria:

* In this study we will include 60 patients (age ranged from 20 to 40 years) with uterine size less than 12 weeks and cavity depth less than 12cm. Different types of intrauterine lesions (submucous fibroids of types 0, 1 and 2 with diameter less than 4 cm, polyps,septum and adhesions).

Exclusion Criteria:

* Any case with the following diseases will be excluded from the study.
* Cardiac diseases (myocardial ischemia, myocardial infarction or valve lesions).
* Renal impairment.
* Neurological affection.
* Chest diseases.
* Hepatic impairment.
* coagulation abnormalities.
* Patient refusal.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — FEMALE IN THE REPRODUCTIVE AGE (20-40 YEARS)
Enrollment: 60 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure | data will be collected over 24 hours from the beginning of the procedure
  Non-invasive blood pressure measurement by using sphygmomanometer cuff

CONTACTS AND LOCATIONS:
Overall Officials: AHMED sonbaty, doctor, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt